CLINICAL TRIAL: NCT02590965
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Phase II Clinical Trial to Evaluate the Efficacy and Safety of Fruquintinib Plus Best Supportive Care in Patients With Advanced Non-squamous Non-small Cell Lung Cancer
Brief Title: A Clinical Trial of Fruquintinib in Patients With Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Collaborators: Shanghai Chest Hospital (Other)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-013-00CH1
Record Dates: First submitted 2015-03-26; First posted 2015-10-29 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — HMPL-013

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Placebo Comparator): Placebo is a capsule in the form of 1mg and 5 mg, orally, once daily, 3 weeks on/1week off with best supportive care.
  Interventions: Drug: Placebo
- Treatment Group (Experimental): The subjects will receive oral Fruquintinib at fasting state 5mg+best supportive care, once daily for the first 3 consecutive weeks and dose holiday for 1 week according to their dose regimens until the occurrence of disease progression, unacceptable toxicity, or withdrawal of consent
  Interventions: Drug: Fruquintinib

INTERVENTIONS:
Drug: Fruquintinib — After checking eligibility criteria, subjects will be randomized into Fruquintinib plus best supportive care group (treatment group) or placebo plus best supportive care group (control group) in a ration of 2:1.
  Other Names: HMPL-013
  Arms: Treatment Group
Drug: Placebo — Placebo is a capsule in the form of 1mg and 5mg, orally, once daily, 3 weeks on/1 week off
  Other Names: HMPL-013-placebo
  Arms: Control Group

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multi-center Phase II clinical trial to evaluate the efficacy and safety of Fruquintinib plus best supportive care in patients with advanced non-squamous non-small cell lung cancer who failed to second-line standard chemotherapy.

DETAILED DESCRIPTION:
Approximately 90 subjects will be randomized to Fruquintinib plus best supportive care or placebo plus best supportive care at a 2:1 ratio.

Randomization will be stratified by EGFR (epidermal growth factor receptor) gene status: mutant vs. wild type vs. unknown.

All subjects will receive Fruquintinib/placebo for consecutive 3 weeks, followed by one-week rest. A treatment cycle consists of 4 weeks. Tumor assessment will be performed every 4 weeks in the first 3 cycles, and every 8 weeks since the 4th cycle, until disease progression. Further treatment and survival follow-up after progression will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the study and sign the informed consent form voluntarily;
2. Histologically and/or cytologically diagnosed with local advanced and/or metastatic stage IIIB/IV non-squamous NSCLC;
3. Previously failed to two chemotherapy regimens(treatment failure is defined as disease progression or intolerable toxicity), patients with positive EGFR mutation permitted to treated by EGFR-TKI previously; patients with EGFR wild type or unknown whether or not treated by EGFR-TKI previously;
4. Aged 18-75 years (inclusive);
5. Body weight ≥40 kg;
6. Evident measurable lesion(s) (according to RECIST1.1);
7. ECOG Performance Status 0-1;
8. Expected survival >12 weeks

Exclusion Criteria:

1. Treatment in another clinical trials in the past 3 weeks; or treatment with systemic anti-tumor chemotherapy, radiotherapy or biotherapy within 3 weeks prior to administration of the study drug;
2. Previous therapy with VEGF/VEGFR inhibitors;
3. Unrecovered from toxicity caused by previous anti-cancer treatment (CTCAE >grade 1), or not completely recovered from previous surgery;
4. Previous active brain metastasis (without radiotherapy previously, or symptoms stable < 4 weeks, or with clinical symptoms, or with medication to control symptoms);
5. Other malignancies except basal cell carcinoma or cervical carcinoma in situ in the past 5 years;
6. Uncontrolled clinical active infection, e.g. acute pneumonia and active hepatitis B;
7. Dysphagia or known drug malabsorption;
8. Present active duodenal ulcer, ulcerative colitis, intestinal obstruction and other gastrointestinal diseases or other conditions that may lead to gastrointestinal bleeding or perforation according to the investigators' judgment; or with a history of intestinal perforation or intestinal fistula;
9. Have evidence or a history of thrombosis or bleeding tendency, regardless of seriousness;
10. Stroke and/or transient ischemic attack within 12 months prior to enrollment;
11. Appropriate organ function. Patients with any of the following conditions will be excluded:

    * Absolute neutrophil count (ANC) <1.5×109/L, platelet <100×109/L or hemoglobin <9 g/dL within 1 week prior to enrollment;
    * Serum total bilirubin >1.5 upper limit of normal (ULN), alanine transaminase and aspartate transferase >1.5×ULN; ALT and AST > 3×ULN in patients with liver metastasis;
    * Electrolyte abnormality of clinical significance;
    * Blood creatinine >ULN and creatinine clearance <60 ml/min;
    * Urine protein 2+ or above, or 24 h urine protein quantification ≥1.0 g/24 h;
    * Activated partial thromboplastin time (APTT) or/and INR and prothrombin time (PT) >1.5×ULN (according to reference range in each clinical study center);
12. Uncontrolled hypertension, systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg with medication; or heart failure NYHA classification ≥ grade 2;
13. Heart function evaluation: left ventricular ejection fraction <50% (echocardiography);
14. Acute myocardial infarction, severe/unstable angina or coronary bypass surgery within 6 months prior to enrollment; history of arterial thrombosis or deep venous thrombosis;
15. Skin wound, surgical site, wound site, severe mucosal ulcer or fracture without complete healing;
16. Female subjects who are pregnant or lactating or of child bearing potential with positive pregnancy test result before the first dose;
17. Patients with child bearing potential who or whose sexual partners are not willing to take contraceptive measures;
18. Any clinical or laboratory abnormalities unfit to participate in this clinical trial according to the investigator's judgment;
19. Serious psychological or psychiatric disorders which may affect subject compliance in this clinical study;
20. Allergy to Fruquintinib and/or excipient contained in trial drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2014-05-29 (Actual); Primary Completion 2015-08-07 (Actual); Study Completion 2017-02-10 (Actual)

PRIMARY OUTCOMES:
Progressive free survival (PFS) | measured every 4 weeks at first 2 cycles and every 8 weeks since the third cycle from randomization to disease progression, assessed up to one year
  To compare the Progressive Free Survival (PFS) of Fruquintinib plus best supportive care (BSC) versus placebo plus BSC in patients advanced non-squamous NSCLC patients who failed to standard second-line chemotherapy according to RECIST 1.1

SECONDARY OUTCOMES:
Objective response rate (ORR) | measured every 4 weeks at first 2 cycles and every 8 weeks since the third cycle from randomization to disease progression, assessed up to one year
  To evaluate objective response rate (ORR) in the two groups according to RECIST 1.1
Disease control rate (DCR) | measured every 4 weeks at first 2 cycles and every 8 weeks since the third cycle from randomization to disease progression, assessed up to one year
  To evaluate disease control rate (DCR) in the two groups according to RECIST 1.1
Overall survival (OS) | every 2 months from randomization to death, assessed up to one year
  To evaluate overall survival (OS) in the two groups
safety and tolerability by incidence, severity and outcome of adverse events | From randomization to 30 days after last dose
  To evaluate the safety and tolerability in the two groups by incidence, severity and outcomes of AEs and categorized by severity in accordance with the NCI CTC AE Version 4.0.

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - 307 Hospital of PLA, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital, Beijing, Beijing Municipality
  - Xi Nan Hospital, Third Military Medical University, Chongqing, Chongqing Municipality
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Linyi Tumor Hospital, Linyi, Shandong
  - The Cancer Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Chengdu, Sichuan
  - The First Affiliated Hosptial of College of Medicine, Zhejiang University, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Lu S, Chang J, Liu X, Shi J, Lu Y, Li W, Yang JJ, Zhou J, Wang J, An T, Yang L, Liu Z, Zhou X, Chen M, Hua Y, Su W. Randomized, Double-Blind, Placebo-Controlled, Multicenter Phase II Study of Fruquintinib After Two Prior Chemotherapy Regimens in Chinese Patients With Advanced Nonsquamous Non-Small-Cell Lung Cancer. J Clin Oncol. 2018 Apr 20;36(12):1207-1217. doi: 10.1200/JCO.2017.76.7145. Epub 2018 Mar 12. PMID 29528793